CLINICAL TRIAL: NCT03490721
Title: Effects of Clustering Care on the Physiological Stability of Preterm Infants in a Neonatal Intensive Care Unit.
Brief Title: Effects of Clustering Care on the Physiological Stability of Preterm Infants.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Abril Nicole Fernandez Oviedo, Principal investigator, Université de Montréal
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Etude_maitrise_2018
Record Dates: First submitted 2018-03-23; First posted 2018-04-06 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Premature Baby 26 to 32 Weeks

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Clustering care for 20 minutes.
  Interventions: Other: Clustering care
- Control (No Intervention): Standard care non clustered.

INTERVENTIONS:
Other: Clustering care — During 20 minutes, preterm infants will receive a cluster care with 2 minutes of hand containment.
  Arms: Intervention

SUMMARY:
This crossover design experimental study aims to compare the physiological stability of premature newborns during and after a cluster of care compared to a period when they receive standard non clustered care at the neonatal unit.

DETAILED DESCRIPTION:
The cluster care will take place at the time of feeding of the premature infants. The intervention will start with a calm period of 20 minutes before the start of care (no manipulations will be allowed), the baby will then received the cluster care for 20 minutes and a quiet period of 30 minutes will follow after the cluster care.

ELIGIBILITY:
Inclusion Criteria:

* between 26 to 31 6/7 weeks of gestation at birth
* more than 72 hours of life,
* receive a respiratory aid such as endotracheal tube, NIPPV (non invasive positive pressures ventilation), CPAP (continuous positive airway pressure) or nasal prongs with oxygen,
* are fed intravenously (IV) or by central venous catheter (CVC),
* one of the parents speaks and reads English or French,
* one of the parents is at least 18 years old to sign the consent.

Exclusion Criteria:

* severely ill (necrotizing enterocolitis, septicemia),
* under respiratory assistance or on a high frequency mode,
* having a congenital or cardiac abnormality,
* requiring surgery,
* sedatives or opioids,
* diagnosed with grade II, III or IV intraventricular hemorrhage and / or hydrocephalus,
* have a device for invasive blood pressure,
* having an oxygen requirement of more than 30% to maintain oxygen saturation within the limits indicated by the NICU (neonatal intensive care unit).
* one of the parents is at least 18 years old to sign the consent.

Ages: 26 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Physiological stability (heart rate, respiratory rate and oxygen saturation) | The physiological stability will be measured for 70 minutes.
  The physiological stability will be measured with the SCRIP score. The Stability of the cardiorespiratory system in premature infants is a scale, in which a score of 0 means major physiological instability and a score of 6 means a physiological stability. For every single parameter there's three grades from severe instability (0 points) to minor instability (1 point) to perfect stability (2 points).

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Aita, PhD, Study Director — Université de Montréal
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The results of this project could be made public in a journal or scientific congress.
Supporting Information: CSR
Time Frame: The results of the study will be available when the study is finished.
Access Criteria: The results will be published in a scientific journal.